CLINICAL TRIAL: NCT05400798
Title: A Longitudinal, Multi-Center Safety Study of Autologous Adult Adipose-Derived Regenerative Cell Injection Into Chronic Partial-Thickness Rotator Cuff Tears
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RC-004
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Partial Thickness Rotator Cuff Tear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adipose Derived Regenerative Cells (Experimental): a single injection of adipose-derived regenerative cells (ADRCs) into the partial-thickness rotator cuff tear
  Interventions: Device: Adipose Derived Regenerative Cells
- Corticosteroid (Active Comparator): a single corticosteroid injection into the subacromial space of the index arm
  Interventions: Device: Corticosteroid

INTERVENTIONS:
Device: Adipose Derived Regenerative Cells — single injection of adipose-derived regenerative cells (ADRCs) into the partial-thickness rotator cuff tear
  Arms: Adipose Derived Regenerative Cells
Device: Corticosteroid — a single corticosteroid injection into the associated subacromial space
  Arms: Corticosteroid

SUMMARY:
This is a longitudinal follow-up study of the RC-002 study, in which up to 246 subjects assigned to two randomization arms will be enrolled: an adipose-derived regenerative cell (ADRC) injection arm (ADRC treatment arm) and the SOC corticosteroid injection arm (active control arm). All subjects will be randomly assigned to ADRC treatment or active control arms in a 2:1 ratio and will be followed up for 6 months.

The goal of the RC-004 study is to enroll all patients that were enrolled and treated in RC-002 and follow for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must have completed RC-002.
* 2. Subjects can give appropriate consent.

Exclusion Criteria:

* 1. Subjects who require the use of index arm for ambulation or mobilization via wheelchair, walker, crutches or cane.
* 2. Subjects whose pain behavior or pain medication usage is, in the opinion of the Investigator, out of proportion to the underlying clinical condition or could interfere with the study-required assessments.
* 3. Subject is on an active regimen of chemotherapy or radiation-based treatment.
* 4. Subject is part of a vulnerable population who, in the judgment of the Investigator, is unable to give informed consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with a mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.
* 5. Uncooperative subjects or those with neurological/psychiatric disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint- Safety | 12 months
  Incidence (%) severity and seriousness of adverse events (AEs)
Primary Endpoint- Safety | 12 months
  Incidence (%) of treatment-related adverse events

SECONDARY OUTCOMES:
Percentage of subjects who demonstrate ≥ 14 mm improvement in VAS - Pain score compared to baseline | 12 months
Percentage of subjects who demonstrate improvement or no worsening of supraspinatus strength on the MRC Muscle Scale compared to baseline | 12 months
Mean improvement in VAS - Pain score compared to baseline | 12 months
Mean improvement in WORC score compared to baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Alt, MD, Study Director — InGeneron, Inc.
Locations (11):
- United States (11):
  - Arizona Research Center, Phoenix, Arizona
  - Biosolutions Clinical Research Center, La Mesa, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Sports and Orthopedic Center, Coral Springs, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Andrews Institute for Orthopedics and Sports Medicine, Gulf Breeze, Florida
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Sanford Orthopedic Clinic/Research, Sioux Falls, South Dakota
  - HD Research, Houston, Texas
  - Texas Center for Cell Therapy and Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No